CLINICAL TRIAL: NCT02500758
Title: Effectiveness of Preoperative Surgical Scrubbing in Reducing Bacterial Load, Using Chlorhexidine Digluconate (CHX) and Parachlorometaxylenol (PCMX)
Brief Title: Effectiveness of Preoperative Surgical Scrubbing Using Clorhexidine Digluconate and Parachlorometaxylenol (ECP)
Acronym: ECP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo Becerro de Bengoa Vallejo (Other)
Responsible Party: Sponsor-Investigator, Ricardo Becerro de Bengoa Vallejo, Doctor of Podiatric Medicine, Universidad Complutense de Madrid
Organization: Universidad Complutense de Madrid (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RBLM
Record Dates: First submitted 2015-06-20; First posted 2015-07-16 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Skin Diseases; Surgical Site Infection
Keywords: Surgical scrubbing; Chlorhexidine digluconate; Parachlorometaxylenol
MeSH Terms: conditions — Skin Diseases; Surgical Wound Infection | interventions — chloroxylenol; Chromogranins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parachlorometaxylenol (Experimental): Reducing bacterial load after preoperative surgical scrubbing using 3% PCMX. Both hands have been prepared by preparatory handwash.
  Interventions: Procedure: Preparatory handwash; Procedure: Preoperative surgical scrubbing using 3% PCMX
- Clorhexidine digluconate (Active Comparator): Reducing bacterial load after preoperative surgical scrubbing using 4% CHG. Both hands have been prepared by preparatory handwash.
  Interventions: Procedure: Preparatory handwash; Procedure: Preoperative surgical scrubbing using 4% CHG

INTERVENTIONS:
Procedure: Preparatory handwash — Preparatory handwash follows the UNE-EN 12791 standard using a diluted soft soap, 200g/1000g, made in community pharmacy service and sterilize in autoclave. Washing hands were prepared without use of a brush for 1 minute with 10 ml of soft soap. After being rinsed with running tap water, they are thoroughly dried with paper towels.
Procedure: Preoperative surgical scrubbing using 3% PCMX — Both hands were scrubbed using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side. The bristled side was used to scrub the entire hands, including all nails, palm and back of the hand, and interdigital spaces, and the foam side was used to rub between the fingers. Each side of each finger, between fingers and back al palm of the hand were rubbed for two and a half minute. Then, the forearms were rubbed from the wrist to the elbow, maintaining the hand highest than the arm, using a minute to wash each side. Both hands were rinsed by current water in an one-way (from the fingertips to the elbow), and wiped with a sterile disposable towel, including nails and interdigital spaces.
  Other Names: Parachlorometaxylenol
  Arms: Parachlorometaxylenol
Procedure: Preoperative surgical scrubbing using 4% CHG — Both hands were scrubbed using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side. The bristled side was used to scrub the entire hands, including all nails, palm and back of the hand, and interdigital spaces, and the foam side was used to rub between the fingers. Each side of each finger, between fingers and back al palm of the hand were rubbed for two and a half minute. Then, the forearms were rubbed from the wrist to the elbow, maintaining the hand highest than the arm, using a minute to wash each side. Both hands were rinsed by current water in an one-way (from the fingertips to the elbow), and wiped with a sterile disposable towel, including nails and interdigital spaces.
  Other Names: Chlorexidine digluconate
  Arms: Clorhexidine digluconate

SUMMARY:
Despite the wide variety of products and antiseptic agents, no agent is ideal for every situation. The investigators would like to evaluate the difference in reducing bacterial load, using 4% chlorhexidine digluconate and 3% parachlorometaxylenol after a preoperative surgical scrubbing.

DETAILED DESCRIPTION:
The investigators conducted a controlled, prospective, randomized study to evaluate the antiseptic effectiveness of preoperative surgical scrubbing using 4% chlorhexidine digluconate and 3% parachlorometaxylenol. Samples were taken from the hands of each volunteer after a preparatory handwash, pre-surgical scrubbing, post-surgical scrubbing and 3 hours after surgical scrubbing.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases.
* Healthy skin on hands, without cuts or abrasions.
* Short and clean fingernails.
* No use of substances with antimicrobial action (e.g. medicated soaps or creams).

Exclusion Criteria:

* History of eczema.
* History of psoriasis.
* Allergies to any of the ingredients of the solutions or contraindication to its use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Becerro de Bengoa Vallejo, DPM, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Becerro de Bengoa Vallejo R, Losa Iglesias ME, Cervera LA, Fernandez DS, Prieto JP. Efficacy of intraoperative surgical irrigation with polihexanide and nitrofurazone in reducing bacterial load after nail removal surgery. J Am Acad Dermatol. 2011 Feb;64(2):328-35. doi: 10.1016/j.jaad.2010.01.011. Epub 2010 Nov 26. PMID 21112671
- [Derived] Vallejo RBB, Fernandez DS, Cervera LA, Aragon LM, Iglesias MEL, Yurrita LRC, Lopez DL. Effectiveness of surgical hand antisepsis using chlorhexidine digluconate and parachlorometaxylenol hand scrub: Cross-over trial. Medicine (Baltimore). 2018 Oct;97(42):e12831. doi: 10.1097/MD.0000000000012831. PMID 30334981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process started in june 2015 and ended in august 2015, involving 20 healthy adult volunteers, who were recruited in Nursing, Physiotherapy and Podiatry School of Complutense University of Madrid.
Pre-assignment Details: The volunteers are randomly divided into two groups of the same size, by tossing a coin.
Groups:
- Parachlorometaxylenol Then Clorhexidine Digluconate: Participants first scrubbed their hands, for 2 minutes, using a sterile disponsable surgical scrub with parachlorometaxylenol After a washout period of 1 week, to allow reconstruction of the normal skin flora, they then scubbed their hands, for 2 minutes, using a sterile disponsable surgical scrub with chlorhexidine digluconato (matching parachlorometaxylenol).
- Chlorhexidine Digluconate Then Parachlorometaxylenol: Participants first scrubbed their hands, for 2 minutes, using a sterile disponsable surgical scrub with chlorhexidine digluconato (matching parachlorometaxylenol).
  After a washout period of 1 week, to allow reconstruction of the normal skin flora, they then scubbed their hands, for 2 minutes, using a sterile disponsable surgical scrub with parachlorometaxylenol.
Period: First Intervention (2 Minutes)
Arm/Group | Parachlorometaxylenol Then Clorhexidine Digluconate | Chlorhexidine Digluconate Then Parachlorometaxylenol
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (1 Week)
Arm/Group | Parachlorometaxylenol Then Clorhexidine Digluconate | Chlorhexidine Digluconate Then Parachlorometaxylenol
Started | 15 | 14
Completed | 13 | 12
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: Second Intervention (2 Minutes)
Arm/Group | Parachlorometaxylenol Then Clorhexidine Digluconate | Chlorhexidine Digluconate Then Parachlorometaxylenol
Started | 13 | 12
Completed | 10 | 10
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Parachlorometaxylenol: Reducing bacterial load after preoperative surgical scrubbing using 3% parachlorometaxylenol. Both hands have been prepared by preparatory handwash.
  Both hands were scrubbed using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side. The bristled side was used to scrub the entire hands, including all nails, palm and back of the hand, and interdigital spaces, and the foam side was used to rub between the fingers. Each side of each finger, between fingers and back al palm of the hand were rubbed for two and a half minute. Then, the forearms were rubbed from the wrist to the elbow, maintaining the hand highest than the arm, using a minute to wash each side. Both hands were rinsed by current water in an one-way (from the fingertips to the elbow), and wiped with a sterile disposable towel, including nails and interdigital spaces.
  Preparatory handwash follows the UNE-EN 12791 standard.
- Chlorhexidine Digluconate: Reducing bacterial load after preoperative surgical scrubbing using 4% chlorhexidine digluconate. Both hands have been prepared by preparatory handwash.
  Both hands were scrubbed using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side. The bristled side was used to scrub the entire hands, including all nails, palm and back of the hand, and interdigital spaces, and the foam side was used to rub between the fingers. Each side of each finger, between fingers and back al palm of the hand were rubbed for two and a half minute. Then, the forearms were rubbed from the wrist to the elbow, maintaining the hand highest than the arm, using a minute to wash each side. Both hands were rinsed by current water in an one-way (from the fingertips to the elbow), and wiped with a sterile disposable towel, including nails and interdigital spaces.
  Preparatory handwash follows the UNE-EN 12791 standard.
- Total: Total of all reporting groups
Arm/Group | Parachlorometaxylenol | Chlorhexidine Digluconate | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.02 (2.05) | 24.62 (3.82) | 24.83 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in the Release of Skin Flora From the Hands From Baseline to 5 Minutes After Disinfection by Surgical Scrubbing (Time Frame- "Baseline and 5 Minutes").
Description: Number of colony-forming units (CFU) sampled up to 5 minutes after disinfection by surgical scrubbing using parachlorometaxylenol or clorhexidine digluconate. After surgical scrubbing and drying, the fingertips are rubbed (including that of the thumb) for 1 minute on the base of a Petri dish containing volumes of 1.0 ml and 0.1 ml of undiluted sampling fluid of TSB and 0.1 ml from its 10-1 dilution are plated out for quantitative culture in TSA.
Time Frame: 5 minutes
Measure: Mean (95% Confidence Interval); unit: CFU/ml
Groups:
- Parachlorometaxylenol: Change in bacterial load after preoperative surgical scrubbing using 3% parachlorometaxylenol. Both hands have been prepared by preparatory handwash.
  Both hands were scrubbed using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side. The bristled side was used to scrub the entire hands, including all nails, palm and back of the hand, and interdigital spaces, and the foam side was used to rub between the fingers. Each side of each finger, between fingers and back al palm of the hand were rubbed for two and a half minute. Then, the forearms were rubbed from the wrist to the elbow, maintaining the hand highest than the arm, using a minute to wash each side. Both hands were rinsed by current water in an one-way (from the fingertips to the elbow), and wiped with a sterile disposable towel, including nails and interdigital spaces.
  Preparatory handwash follows the UNE-EN 12791 standard
- Chlorhexidine Digluconate: Change in bacterial load after preoperative surgical scrubbing using 4% chlorhexidine digluconate. Both hands have been prepared by preparatory handwash.
  Both hands were scrubbed using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side. The bristled side was used to scrub the entire hands, including all nails, palm and back of the hand, and interdigital spaces, and the foam side was used to rub between the fingers. Each side of each finger, between fingers and back al palm of the hand were rubbed for two and a half minute. Then, the forearms were rubbed from the wrist to the elbow, maintaining the hand highest than the arm, using a minute to wash each side. Both hands were rinsed by current water in an one-way (from the fingertips to the elbow), and wiped with a sterile disposable towel, including nails and interdigital spaces.
  Preparatory handwash follows the UNE-EN 12791 standard.
Arm/Group | Parachlorometaxylenol | Chlorhexidine Digluconate
Number analyzed (Participants) | 20 | 20
CFU/ml | 3.96 [3.57 to 4.35] | 3.87 [3.29 to 4.45]

2. Secondary Outcome: Change in the Release of Skin Flora From the Hands From Baseline to 3 Hours After Surgical Scrub Disinfection, Wearing Surgical Gloves (Time Frame- "Baseline and 3 Hours").
Description: Number of colony-forming units (CFU) sampled 3 hours after disinfection by surgical scrubbing using parachlorometaxylenol or clorhexidine digluconate, using surgical gloves. After surgical scrubbing, drying and wearing surgical gloves, the fingertips are rubbed (including that of the thumb) for 1 minute on the base of a Petri dish containing volumes of 1.0 ml and 0.1 ml of undiluted sampling fluid of TSB and 0.1 ml from its 10-1 dilution are plated out for quantitative culture in TSA.
Time Frame: 3 hours
Measure: Mean (95% Confidence Interval); unit: CFU/ml
Arm/Group | Parachlorometaxylenol | Chlorhexidine Digluconate
Number analyzed (Participants) | 20 | 20
CFU/ml | 4.54 [3.92 to 5.16] | 4.65 [3.85 to 5.45]

ADVERSE EVENTS:
Time Frame: A week
Arm/Group | Parachlorometaxylenol | Chlorhexidine Digluconate
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No